CLINICAL TRIAL: NCT05459103
Title: The Effectiveness of Remote Interactive Intervention for Loneliness, Quality of Life, and Social Support Among Seniors in Communities During the COVID-19 Pandemic: A Randomized Controlled Experiment
Brief Title: Remote Interactive Intervention for Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Shang-Yu (Other)
Responsible Party: Sponsor-Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Remote interactive
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Older Adults

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group received a 12-week bidirectional remote interaction intervention.
  Interventions: Other: Bidirectional remote interaction intervention
- Control group (Experimental): Participants in the control group received a 12-week unidirectional remote interaction intervention.
  Interventions: Other: Unidirectional remote interaction intervention

INTERVENTIONS:
Other: Bidirectional remote interaction intervention — Intervention group participants engaged in a 12-week bidirectional remote interaction. All interactions were conducted through the same group on Line. A one-hour interactive online group intervention was held every Monday to Friday from 14:30 to 15:30, for a total of 60 hours. The online interactive interventions were conducted in a structured course format, with a facilitator conducting live classes and alternating between static and dynamic classes.
  Arms: Intervention group
Other: Unidirectional remote interaction intervention — Control group participants engaged in a 12-week unidirectional remote interaction. All interactions were conducted through the same group on Line. Research assistants posted a YouTube video on the Line group at 14:30 every day, Monday through Friday, covering art, music, senior sports, long-term care resources, travel, and food preparation.
  Arms: Control group

SUMMARY:
Background:

During the COVID-19 pandemic, governments around the world adopted the practice of physical distancing, which increased the loneliness experienced by seniors and indirectly affected their quality of life and social support. Remote interaction through online social apps may be the safest and easiest way to address these problems. However, the empirical research on this issue is very limited.

Objective:

This study investigated the impact of a 12-week remote interaction intervention on loneliness, quality of life, and social support for seniors living in a community during the COVID-19 pandemic.

Methods:

This study adopted a randomized controlled trial design and was conducted in communities in central Taiwan. Participants in the intervention group received a 12-week bidirectional remote interaction intervention, while participants in the control group received a 12-week unidirectional remote interaction intervention. The study's primary assessment tools were the UCLA Loneliness Scale and the World Health Organization Quality of Life-BREF Scale (WHOQOL-BREF). The secondary assessment tool was the Inventory of Socially Supportive Behavior.

ELIGIBILITY:
Inclusion Criteria:

* Participants had to satisfy several inclusion requirements. They had to (1) be seniors aged 65 years or older; (2) be able to communicate in Mandarin and Taiwanese; (3) have an MMSE score higher than 20 20 (following Chiang et al., 2010); (4) be able to use a smartphone; and (5) have no previous psychiatric diagnosis.

Exclusion Criteria:

* The study excluded (1) those who were unable to understand how to use Line or YouTube; (2) participants in the experimental group who did not fully participate in the 12-week intervention (at least three days of interaction per week); (3) those who were unable to understand the content of the questionnaire or cooperate with those assigned to help them fill it in; and (4) those who had a major illness or surgery such as a fracture within the last three months.

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
UCLA Loneliness Scale (UCLA) | 10-20 minutes
  The third version of UCLA compiled by Russel (1996) was used to measure "loneliness." It was translated into Chinese by Chang and Yang (1999) and included 20 questions. Each question was scored on the 4-point Likert Scale, with 1: "I never feel this way," 2: "I rarely feel this way," 3: "I sometimes feel this way," and 4: "I often feel this way." The total score ranged between 20 and 80, and the higher the score, the higher the participant's degree of loneliness.
WHO Quality of Life-BREF (WHOQOL-BREF) Scale | 10-20 minutes
  The questionnaire was composed of questions on QOL formulated by the World Health Organization (WHO) based on the commonality of various cultures. The Taiwanese version of WHOQOL-BREF included 28 questions, each scored on a 5-point Likert Scale. It was composed of four domains, namely, Physical health (7 questions), Psychological health (6 questions), Social relationships (4 questions), and Environment (9 questions). The score of an individual question ranged between 1 and 5, and after conversion, the total score of each domain ranged between 4 and 20. The higher the score, the higher the individual's QOL.

SECONDARY OUTCOMES:
Inventory of Socially Supportive Behavior (ISSB) Scale | 10-20 minutes
  Initially developed by Barrera Jr et al. (1981), ISSB was subsequently translated into Chinese and compiled into 8 questions by Ou (2013). The scale consisted of two categories, namely Emotional Support and Tangible Support. The total score of both categories represented the participant's satisfaction with social support. The scale was scored on a 5-point Likert Scale, with 1 representing "Strongly disagree," 2: "Disagree," 3: "Neutral," 4: "Agree," and 5: "Strongly agree." The total score ranged between 8 and 40, and the higher the score, the higher the participant's satisfaction with social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan